CLINICAL TRIAL: NCT05838040
Title: General Exercises With and Without TA Contraction in Patients With Nonspecific Acute LBP: A Crossover Randomised Controlled Trial
Brief Title: General Exercises With and Without TA Contraction in Patients With Nonspecific Acute LBP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 012/004221
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General Exercises (Active Comparator): This exercise activates paravertebral and abdominal muscles. Because this exercise impose extra loading on the spinal tissues, the general exercise was selected on the basis of maximizing the contraction benefit/spinal loading ratio.
  Interventions: Other: General exercises
- General exercises with TA contraction (Experimental): This exercise activates paravertebral and abdominal muscles. Because this exercise impose extra loading on the spinal tissues, the general exercise was selected on the basis of maximizing the contraction benefit/spinal loading ratio. The patients will be asked to contract TA will doing these exercises.
  Interventions: Other: General exercises with tranversus abdmoinis contraction

INTERVENTIONS:
Other: General exercises — General exercise is a structured exercise program designed to help individuals with back pain improve their fitness levels. The program comprises of a series of exercise classes that are led by a physiotherapist. The classes involve a combination of aerobic, strength, and flexibility exercises, and aim to improve overall physical fitness, reduce pain, and improve function. The program is specifically designed for individuals with back pain, and the exercises are tailored to meet the needs of each participant. The Back to Fitness Program is based on the principles of exercise prescription and is intended to be a safe and effective way to manage back pain through exercise.
  Arms: General Exercises
Other: General exercises with tranversus abdmoinis contraction — General exercise is a structured exercise program designed to help individuals with back pain improve their fitness levels. The program comprises a series of exercise classes that are led by a physiotherapist. The classes involve a combination of aerobic, strength, and flexibility exercises, and aim to improve overall physical fitness, reduce pain, and improve function. The program is specifically designed for individuals with back pain, and the exercises are tailored to meet the needs of each participant. In addition to these exercises, the Back to Fitness Program includes the activation of the transverse abdominis muscle, which is an important stabilizing muscle in the core. The activation of this muscle is done through specific exercises and techniques, and is intended to improve core stability and reduce the risk of further back injuries.
  Arms: General exercises with TA contraction

SUMMARY:
PURPOSE: To evaluate the effectiveness of adding transversus abdominis contraction to general exercises to treat patients with nonspecific acute low back pain.

BACKGROUND: Non-specific low back pain affects people of all ages and is a leading contributor to disease burden worldwide. Management consists of education and reassurance, analgesic medicines, non-pharmacological therapies, and timely review. The clinical course of low back pain is often favourable; thus, many patients require little if any formal medical care. Two treatment strategies are currently used, a stepped approach beginning with more simple care that is progressed if the patient does not respond, and the use of simple risk prediction methods to individualise the amount and type of care provided. Motor control exercises, which advocate the contraction of the TrA have shown some efficacy for patients with chronic low back pain. However, the validity of this strategy for patients with acute LBP is unclear.

HYPOTHESES: there will be no significant effect of adding transversus abdominis contraction to general exercise than general exercise alone in patients with non-specific acute low back pain.

RESEARCH QUESTION: Is there a statistically significant effect of adding transversus abdominis contraction to general exercise on outcomes of patients with non-specific acute low back pain?

ELIGIBILITY:
Inclusion Criteria:

1. Individuals of both sexes
2. Aged between 18 and 50 years
3. Acute nonspecific low back pain according to The most recent guidelines for the diagnosis and management of NSLBP come from the American College of Physicians and were published in 2017. According to these guidelines, the diagnosis of acute NSLBP should be made based on the following criteria:

Acute onset of low back pain, defined as pain lasting for less than 12 weeks No specific identifiable cause of the pain (e.g., infection, malignancy, fracture, inflammatory disorder) No radicular symptoms (e.g., pain radiating down the leg) No significant neurological deficits or findings on physical examination (e.g., loss of reflexes or muscle strength)

Exclusion Criteria:

1. Serious low back pathology
2. Contraindications to exercise therapy
3. Neurological signs (leg weakness)
4. Specific spinal pathology (e.g., malignancy, or inflammatory joint or bone disease)
5. Prior back surgery

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-21 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity via numeric pain rating scale | Changes in pain intensity at baseline, 10 weeks after randomization, 3 and 6 months after discharge.
  The primary outcome measure is pain intensity, which will be assessed using a numeric pain rating scale. Participants will be asked to rate their pain intensity on a scale of 0 to 10, with 0 indicating no pain and 10 indicating the worst possible pain. Pain intensity will be measured at four time points: baseline, 10 weeks after randomization, 3 months after discharge, and 6 months after discharge. The change in pain intensity from baseline to each follow-up time point will be analyzed using appropriate statistical methods. The primary objective of the study is to determine whether the Back to Fitness Program is effective in reducing pain intensity over time.

SECONDARY OUTCOMES:
Pain Pressure Threshold | Changes at Pain pressure threshold at baseline, 10 weeks after randomization, 3 and 6 months after discharge.
  Pain pressure threshold is a measure of the minimum amount of pressure that causes pain in the affected area. It will be assessed using a pressure algometer.
Disability | Changes in Disability at baseline, 10 weeks after randomization, 3 months after discharge, and 6 months after discharge.
  Disability will be assessed using the Roland-Morris Disability Questionnaire, which is a self-reported questionnaire that assesses the impact of back pain on daily activities. The questionnaire includes 24 items that ask participants to rate their ability to perform various activities on a scale of 0 to 24. Higher scores indicate greater disability.
Global Perception Effect | changes in Global perception at baseline, 10 weeks after randomization, 3 months after discharge, and 6 months after discharge.
  Global perception effect is a measure of the participant's overall perception of the effectiveness of the general exercise in reducing pain and improving function. It will be assessed using a single-item question that asks participants to rate their perception of the program's effectiveness on a scale of 0 to 10. Higher scores indicate greater effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Chair — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) collected during this study will be available upon reasonable request. Requests for access to the data should be submitted via email to mohamed.elmeligie@acu.edu.eg. All requests will be reviewed by the study investigators to ensure that they are reasonable and consistent with the ethical principles of the study. Access to the data will be granted in compliance with applicable laws and regulations, and with appropriate safeguards to protect the privacy and confidentiality of study participants.
Supporting Information: SAP, ICF, CSR
Time Frame: During the trial and after 1 year of the end of trial.
Access Criteria: via email to mohamed.elmeligie@acu.edu.eg